CLINICAL TRIAL: NCT00004738
Title: Genetic Analysis of the Chiari I Malformation
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000089; 00-N-0089
Record Dates: First submitted 2000-02-26; First posted 2000-02-28 (Estimated); Last update posted 2026-01-26 (Actual); Status verified 2026-01-22

CONDITIONS: Syringomyelia; Type I Arnold Chiari Malformation
Keywords: Arnold Chiari Malformation; Skeletal Dysplasia; Syringomyelia; Genetics; Natural History
MeSH Terms: conditions — Syringomyelia; Arnold-Chiari Malformation; Mucopolysaccharidosis IV

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Family Members: At least 2 family members of a patient with a confirmed diagnosis of Chiari I malformation.
- Patients: Patient with a confirmed diagnosis of Chiari I malformation who has a family member with syringomyelia or Chiari I malformation

SUMMARY:
The purpose of this study is to better understand the genetic factors related to the Chiari I malformation. In people with this abnormality, the lower part of the skull is smaller than normal. As a result, the lowest part of the brain, called the cerebellar tonsils, protrudes out of the hole at the bottom of the skull into the spinal canal. This study will try to discover the location of the genes responsible for the malformation.

Candidates for this study are: 1) Patients with Chiari I malformation who also have a family member with the abnormality or a family member with syringomyelia (a cyst in the spinal cord that is often associated with the Chiari I malformation). 2) Family members of patients with the Chiari I malformation.

Participants will have a medical history and physical and neurologic examinations. They will undergo magnetic resonance imaging (MRI) of the brain and cervical (neck) spinal cord to measure the size of the head and determine the presence of the Chiari I malformation and syringomyelia. A small blood sample (about 2 tablespoons) will be drawn for DNA studies relating to the Chiari I malformation.

DETAILED DESCRIPTION:
Objectives: The goal of this study is to establish family pedigrees and undertake genetic linkage analysis that will identify gene loci associated with the Chiari I malformation and underdevelopment of the bone forming the posterior cranial fossa.

Study Population: Patients and family members of patients with the Chiari I malformation. Because the research institutions are located in the United States and Russia, subjects will be recruited predominantly from these countries.

Design: Human subjects will undergo 1) neurologic examinations, 2) head and cervical MRI scans to evaluate for the Chiari I malformation, syringomyelia, and maldevelopment of the posterior fossa, and 3) isolation and analysis of genomic DNA from whole blood for linkage analysis.

Outcome Measures: Pedigrees will be established based on the MRI findings. The Chiari I phenotype will be defined as the caudal portion of the cerebellar tonsils lying greater than or equal to 2 mm below the foramen magnum and underdevelopment of the bone of the posterior fossa will be defined as 1) obliteration of the CSF pathways in the inferior portion of the posterior fossa, 2) posterior fossa volume to supratentorial volume ratio of less than or equal to 15%, or 3) abnormal shortening of the bones of the skull base. Genetic analysis of the genomic DNA will be performed with DNA polymorphic markers to identify chromosomal loci linked to the small posterior fossa phenotype. A lod score of 3.0 (equivalent to 1000:1 odds in favor of linkage) will be taken as proof that the Chiari I gene maps to the same genetic region of the human genome as a given DNA marker.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible for entry into the study, a candidate must meet the following criteria:

Patient with a confirmed diagnosis of Chiari I malformation who has a family member with syringomyelia or Chiari I malformation, or

Family member of a patient with a confirmed diagnosis of Chiari I malformation, AND

There are at least two family members diagnosed with Chiari I malformation.

If an adult, able to give informed consent; if a minor, has an adult who is legally responsible for the subject and who is able to give consent.

EXCLUSION CRITERIA:

A candidate will be excluded if he/she:

Has a contraindication to MRI scanning.

Is unable to comprehend the risks of the testing.

Is less than one year of age.

Cannot undergo MRI scanning without sedation.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with a confirmed diagnosis of Chiari I malformation who has a family member with syringomyelia or Chiari I malformation, or family member of a patient with a confirmed diagnosis of Chiari I malformation.
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2001-06-04 (Actual)

PRIMARY OUTCOMES:
Family Pedigree/Genetic Linkage | ongoing
  Establish family pedigrees and undertake genetic linkage analysis that will identify gene loci associated with the Chiari I malformation andunderdevelopment of the bone forming the posterior cranial fossa.
Genetic Analysis | Genetic Analysis ongoing
  Genetic analysis of the genomic DNA will be performed with DNA polymorphic markers to identify chromosomal loci linked to the Chiari I and small posterior fossa phenotype.

CONTACTS AND LOCATIONS:
Overall Officials: John D Heiss, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (2):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States
- Kazan State Medical University, Kazan', Russia

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2000-N-0089.html